CLINICAL TRIAL: NCT00820599
Title: Transfemoral Placement of AoRtic Balloon Expandable Transcatheter VAlves TrIaL (EUROPE)
Brief Title: PREVAIL-TF: Transfemoral Placement of Aortic Balloon Expandable Transcatheter Valves Trial (Europe)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-04
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Aortic Valve Stenosis
Keywords: Sapien Valve; Cardiovascular Diseases; Valvular Heart Disease; Aortic Stenosis; Heart Valve Therapy; Transfemoral; Transcatheter
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVR (Experimental): Transaortic Valve Replacement
  Interventions: Device: Sapien XT™ transcatheter heart valve and delivery system

INTERVENTIONS:
Device: Sapien XT™ transcatheter heart valve and delivery system

SUMMARY:
A single arm, prospective multicenter non-randomized confirmatory clinical trial evaluating the Edwards SAPIEN XT™ transcatheter heart valve (model 9300TFX; "study valve"), its transfemoral delivery system, and crimper accessories. The trial includes a premarket confirmatory cohort to evaluate the system performance as well as a Post Market Clinical Follow-up phase involving expanded enrollment and long-term follow-up of all patients to evaluate valve performance out to 5 years.

DETAILED DESCRIPTION:
Edwards Lifesciences obtained CE marking authorization for transfemoral delivery / implantation of the Edwards SAPIEN™ transcatheter heart valve (model 9000TFX) using the RetroFlex™ delivery system in August 2007 and introduced these devices for commercial distribution in the European Economic Area (EEA) in October 2007.

Clinical Sites: Up to 11 sites in Europe

ELIGIBILITY:
Inclusion Criteria:

All candidates for this study must meet all of the following inclusion criteria:

1. Patients must have co-morbidities such that the surgeon (Co Investigator) and interventional cardiologist (Principal Investigator) concur that the predicted risk of operative mortality is > 15% with a minimum STS Risk Calculator score of ≥ 10 and/or Logistic EuroSCORE of > 20%.
2. Patient is symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class II or greater.
3. The subject or the subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided a written informed consent that has been approved by the reviewing Ethics Committee (EC) of the respective clinical site.
4. Subject is willing to comply with specified follow up evaluations, including possible coronary angiography and transesophageal echocardiography.
5. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

Exclusion Criteria:

1. Aortic valve is a congenital unicuspid or bicuspid valve, or is non-calcified.
2. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).
3. Any therapeutic invasive cardiac procedure, other than BAV, performed within 30 days of the index procedure (or 6 months if the procedure was a drug eluting coronary stent implantation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Stefan Sack, Study Director — Cardiology Clinic of Schwabing Clinic; Isabelle Fourthin, Study Director — Edwards Lifesciences SA
Locations (11):
- Ornze Lieve Vrouwziekenhuis (OLVZ) Aalst, Aalst, Belgium
- France (4):
  - Institut Hospitalier Jacques Cartier, Massy
  - Hospital Bichat Claude Bernard, Paris
  - CHU Hospital Charles Nicolle, Rouen
  - Clinique Pasteur, Toulouse
- Germany (4):
  - Hamburg University Cardiovascular Center, Hamburg
  - City Clinics Karlsruhe, Karlsruhe
  - Heart Center Leipzig, Leipzig
  - Schwabing Clinic, Munich
- United Kingdom (2):
  - St. Thomas' Hospital - NHS Trust, London
  - Kings College Hospital - NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One patient withdrew prior to procedure. Prior to procedure, two patients were noted as having significant co-morbidities not accounted for by the Euroscore, therefore they were exited from the trial prior to procedure.
Pre-assignment Details: Three enrolled subjects did not enter the procedure room.
Groups:
- TAVR: Transaortic Valve Replacement
  Sapien XT™ transcatheter heart valve and delivery system
Period: Overall Study
Arm/Group | TAVR
Started | 211
Completed | 80
Not Completed | 131
Not completed — Death | 129
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | TAVR
Number analyzed (Participants) | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 83.2 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 69
STS Risk Score [Mean (Standard Deviation); unit: Units on Scale] — The Society of Thoracic Surgeons (STS) Score measures patient risk of mortality or morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk of operative mortality.
  Units on Scale | 9.1 (6.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Deaths
Description: Number of death at 30-days from the index procedure.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR
Number analyzed (Participants) | 211
Participants | 21

2. Secondary Outcome: Number of Participants With a Stroke
Description: Total number of participates with a stroke.
Time Frame: 30 days from the index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR
Number analyzed (Participants) | 211
Participants | 9

ADVERSE EVENTS:
Time Frame: 5 Years
Arm/Group | TAVR
All-Cause Mortality (participants affected / at risk) | 129/211
Serious Adverse Events (participants affected / at risk) | 193/211
Other Adverse Events (participants affected / at risk) | 192/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR (N=211)
Aneurysm (Vascular disorders) | 1 (1)
Angina (Cardiac disorders) | 11 (16)
Annular Dissection (Injury, poisoning and procedural complications) | 2 (2)
Aortic Dissection (Vascular disorders) | 1 (1)
Aortic Regurgitation ( 3+ 0r 4+) (Cardiac disorders) | 2 (2)
Arrhythmia and Pacemaker Implant (Cardiac disorders) | 31 (31)
Arrhythmia w/o Pacemaker Implant (Cardiac disorders) | 20 (23)
Bleeding Event Major - Not Surgical (Vascular disorders) | 19 (22)
Bleeding Event Minor - Not Surgical (Vascular disorders) | 18 (18)
Bone Fracture (Injury, poisoning and procedural complications) | 24 (26)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (20)
Cardiac Tamponade (Cardiac disorders) | 5 (5)
Circulatory Disorders (Cardiac disorders) | 3 (4)
Coagulopathy / Hematological Disorder (Blood and lymphatic system disorders) | 27 (31)
Death (General disorders) | 130 (130)
Drug Reaction (General disorders) | 1 (1)
Embolism - Not Stroke - Not TE (Vascular disorders) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2)
Explant (Surgical and medical procedures) | 3 (3)
Fever Unknown Origin (General disorders) | 3 (3)
Gastro-Intestinal Compl (Gastrointestinal disorders) | 15 (23)
Heart Failure (Cardiac disorders) | 70 (123)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 4 (4)
Infection / Inflammation (Infections and infestations) | 45 (61)
Metabolic Complication (Metabolism and nutrition disorders) | 8 (8)
Mitral Regurg. ( 3+ or 4+) (Cardiac disorders) | 1 (1)
Multiple Organ Comp/Failure (General disorders) | 18 (18)
Myocardial Damage (Injury, poisoning and procedural complications) | 4 (4)
Myocardial Infarction (Cardiac disorders) | 16 (18)
Neurological Event Minor - Not Stroke (Nervous system disorders) | 12 (13)
Neurological Event Severe - Not Stroke (Nervous system disorders) | 1 (1)
Other (General disorders) | 57 (95)
Pericardial Effusion (Cardiac disorders) | 7 (7)
Peripheral Edema (General disorders) | 1 (1)
Perivalvular Leak (1+ or 2+) (Product Issues) | 1 (1)
Perivalvular Leak (3+ or 4+) (Product Issues) | 7 (7)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Renal Comp / Failure Not Requiring Dialysis (Renal and urinary disorders) | 18 (20)
Renal Failure Requiring Dialysis (Renal and urinary disorders) | 12 (13)
Reoperation (Surgical and medical procedures) | 5 (5)
Respiratory Comp / Failure (Respiratory, thoracic and mediastinal disorders) | 28 (38)
Sepsis (Infections and infestations) | 10 (10)
Stroke - Bleeding Origin (Nervous system disorders) | 1 (1)
Stroke - Embolic Origin (Nervous system disorders) | 10 (10)
Stroke - Unknown Origin (Nervous system disorders) | 5 (5)
Sudden Death (General disorders) | 19 (19)
Suicide (Psychiatric disorders) | 1 (1)
Surgical Bleeding (Injury, poisoning and procedural complications) | 9 (9)
Syncope (Nervous system disorders) | 9 (12)
Thromboembolic Event Minor - Not Stroke (Vascular disorders) | 1 (1)
Thrombus (Vascular disorders) | 1 (1)
Transitory Psychotic Syndrome (Psychiatric disorders) | 2 (2)
Tricuspid Regurg. ( 3+ or 4+) (Cardiac disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 5 (6)
Valve Embolization (General disorders) | 1 (1)
Valve Malpositioned (Injury, poisoning and procedural complications) | 3 (3)
Valve Migration (Product Issues) | 2 (2)
Vascular Access-Related Complication (Injury, poisoning and procedural complications) | 24 (26)
Vascular Complication (Not Access-Related) (Vascular disorders) | 13 (32)
Vision Disorder (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR (N=211)
Arrhythmia w/o Pacemaker Implant (Cardiac disorders) | 58 (66)
Bleeding Event Minor - Not Surgical (Vascular disorders) | 42 (49)
Coagulopathy / Hematological Disorder (Blood and lymphatic system disorders) | 51 (58)
Ecg Changes (Cardiac disorders) | 19 (22)
Fever Unknown Origin (General disorders) | 11 (11)
Gastro-Intestinal Compl (Gastrointestinal disorders) | 29 (37)
Heart Failure (Cardiac disorders) | 32 (36)
Hypertension (Vascular disorders) | 16 (19)
Hypotension (Vascular disorders) | 15 (15)
Infection / Inflammation (Infections and infestations) | 72 (93)
Metabolic Complication (Metabolism and nutrition disorders) | 29 (40)
Neurological Event Minor - Not Stroke (Nervous system disorders) | 41 (50)
Other (General disorders) | 105 (217)
Peripheral Edema (General disorders) | 21 (25)
Perivalvular Leak (1+ or 2+) (Product Issues) | 21 (21)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 32 (38)
Renal Comp / Failure Not Requiring Dialysis (Renal and urinary disorders) | 32 (38)
Respiratory Comp / Failure (Respiratory, thoracic and mediastinal disorders) | 21 (23)
Transitory Psychotic Syndrome (Psychiatric disorders) | 19 (20)
Urinary Tract Infection (Infections and infestations) | 25 (36)
Vascular Access-Related Complication (Injury, poisoning and procedural complications) | 29 (33)
Vision Disorder (Eye disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes